CLINICAL TRIAL: NCT05197530
Title: Near InfraRed Fluorescence Imaging of Lymphatic Transport Using Indocyanine Green: Phase II Pilot
Brief Title: Imaging of Lymphatic Vessels in People with Rheumatoid Arthritis (RA)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Christopher Ritchlin, Professor, University of Rochester
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY6830; 2R01AR056702-11A1 (NIH)
Record Dates: First submitted 2022-01-03; First posted 2022-01-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Near InfraRed; Lymphatic Transport; Imaging; Indocyanine Green; ICG; Rheumatoid Arthritis; MSImager
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early RA (<1 year of disease) (Experimental): In this single center study, early RA subjects (<1 year of disease) who are MTX inadequate responders or experience a flare (see inclusion criteria for detail) on MTX and are starting an anti-TNF therapy will be invited to participate to receive ICG injections at Baseline (prior to the start of medication), week 16 and week 52. NIR-ICG imaging will be done immediately post injection and 1 week later for a total of three injection/imaging visits and three imaging visits without injections. See schedule of events for more detail. Total length of participation will be up to 53 weeks (+3days).
  Interventions: Drug: Indocyanine green; Device: MultiSpectral Imaging System
- Established RA (> 10 years of disease) (Experimental): Patients with symptomatic established RA (>10 years) will be invited to participate in an ICG injections followed by NIR-ICG imaging and NIR-ICG imaging visit 1 week later. Total length of participation will be up to 1 week (+3 days)
  Interventions: Drug: Indocyanine green; Device: MultiSpectral Imaging System

INTERVENTIONS:
Drug: Indocyanine green — A trained physician will inject 0.1 ml of the ICG in to the web spaces of the hands in both upper extremities.
  Other Names: ICG; IC-Green; 1748-701-02
Device: MultiSpectral Imaging System — Once the ICG is injected, the contrast is expected to fluoresce underneath the MultiSpectral Imaging System. Multispectral video and still images will be recorded at the study visits.
  Other Names: MSImager

SUMMARY:
Lymphatic transport was previously examined by these investigators using Near InfraRed Indocyanine Green fluorescence imaging (NIR-ICG) of the upper extremities. They established reliable and reproducible methodologies in RA patients. The purpose of this phase 2 pilot is to study RA disease progression and effectiveness as well as the mechanism of action of clinical interventions using established NIR-ICG methodologies in previous studies.

DETAILED DESCRIPTION:
In preclinical studies, these investigators demonstrated that amelioration of tumor necrosis factor (TNF)-induced arthritis with anti-TNF, but not methotrexate (MTX) therapy, correlates with normalization of ICG clearance and popliteal lymph node (PLN) contractions. In RA patients during hand flare, it was found that ICG clearance from the web spaces, and numbers of ICG+ lymphatic basilic vessels of RA hands, are significantly decreased vs. healthy controls. Based on these observations, two important questions warrant testing to assess the clinical utility of NIR-ICG biomarkers in RA hands: Does amelioration of active synovitis pre and post treatment) correlate with: 1) increased ICG clearance (primary outcome) and/or 2) recovery of basilic ICG+ vessels (secondary outcome)? To formally address these questions, a clinical pilot will be conducted of early RA patients with symptomatic disease in their hand(s), who will undergo NIR-ICG imaging at baseline, 16-weeks, and 1-year post anti-TNF therapy, and examine if NIR-ICG outcome measures predict and correlate with clinical response.

ELIGIBILITY:
Inclusion Criteria:

Early RA

* Ability to provide written informed consent
* Subjects must be 18 years old or older
* RA subjects must fulfill 2010 American College of Rheumatology (ACR) criteria with a DAS28-C-Reactive Protein (CRP) >3.5
* Must have 1 year or less of disease
* Must be MTX inadequate responder (DAS28-CRP >2.6 at 4 months of therapy) OR experience a flare on MTX (self-reported and score of >25 on the Outcome Measures in Rheumatology (OMERACT) Flare questionnaire AND are starting an anti-TNF therapy.
* Must have active synovitis in one or both hands confirmed by ultrasound

Established RA

* Ability to provide written informed consent
* Subjects must be 18 years of age or older
* RA subjects must fulfill 2010 ACR criteria with a DAS-CRP >3.5
* Must have at least 10 years of disease
* Must have active synovitis in one or both hands confirmed by ultrasound
* Must be on a stable dose of DMARD (MTX, leflunomide, azulfidine, hydroxychloroquine), Janus Kinase (JAK) inhibitor or biologic agent for 8 weeks

Exclusion Criteria: All PATIENTS

* Active systemic disorders or inflammatory conditions other than RA, (i.e., chronic infections with hepatitis B, hepatitis C or HIV) that would confound the study results.
* Known sensitivity to iodine because of residual iodide in Indocyanine Green
* Pregnant women should not participate; pregnancy tests will not be performed
* Inability to donate blood due to poor venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clearance | 1 week post injection
  The change in Indocyanine Green signal intensity (arbitrary units) over time is measured by observing the fluorescence using the Multispectral Imaging System. The MSImager software analyses the signal intensity. This outcome measure will be quantified for both early RA and late RA subjects.

SECONDARY OUTCOMES:
Lymphatic Vessels | 16 weeks
  Using 2D still images from the NIR scanning sessions, lymphatic vessel location will be identified, and vessel numbers will be quantified. Comparisons with 2D images will be performed to identify vessel location and numbers. The images will then be superimposed upon each other in order to confirm concordance of lymphatic vessels. This outcome measure will be quantified for both early RA and late RA subjects.
Contraction Rate | 16 weeks
  The contraction rate is measured as lymphatic vessel contractions/min in the dominant lymphatic vessel efferent to the injection site using the MultiSpectral Imaging System (MSImager) that captures real time movies. The MSImager software analyses the signal intensity to determine the contraction rate. This outcome measure will be quantified for both early RA and late RA subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ritchlin, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States